CLINICAL TRIAL: NCT02221115
Title: A Survey-driven Evaluation of Patients Response to the Introduction of Google Glass in the Orthopaedic Trauma Clinic
Brief Title: A Survey of Google Glass by Orthopaedic Trauma Patients and Surgeons
Acronym: GoogleGlass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Edward Harvey, MDCM FRCSC, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SDR 14.135; RI-MUHC - MGH (Other: RI-MUHC - Montreal General Hospital)
Record Dates: First submitted 2014-07-24; First posted 2014-08-20 (Estimated); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Orthopedic Disorders; Trauma
Keywords: Google Glass device; Evaluation; patient's; response; to new technology; clinical setting
MeSH Terms: conditions — Musculoskeletal Diseases; Wounds and Injuries | interventions — Smart Glasses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Google Glass (Other): Investigators using Google Glass during clinic visit
  Interventions: Device: Google Glass
- No Google Glass (No Intervention): Investigator will not be using Google Glass during clinic visit

INTERVENTIONS:
Device: Google Glass — The device is a wearable, voice-controlled Android device that resembles a pair of eyeglasses and displays information directly in the user's field of vision
  Arms: Google Glass

SUMMARY:
Patients seen in the Orthopaedic Trauma clinic will be asked to consent for potential video/picture recording using the Google Glass device during their visit with the orthopaedic surgeon or resident.

The investigators want to record the patient's level of acceptance and response to this new technology. There are two arms: Patients seen by a doctor wearing the Google Glass device and those that will not be exposed. Both groups will be asked to complete a survey after their clinic visit.

The device users (doctor) will complete a survey which will evaluate how effective this new tool is in the Orthopaedic clinical setting.

DETAILED DESCRIPTION:
Google Glass is a new low-profile wearable technology that allows physicians to record hands-free video and pictures and to directly video link and communicate with other wearers of this device. In addition to this, the device has a heads up display that is capable of searching the internet on voice command. The device has the same functionality as a smart phone with the benefit of being hands-free and wearable. The device is currently in a beta testing period where "Explorers" are accepted by application to a program to use and assess the device. The investigators have been able to obtain three of these devices.

The Google Glass device has the ability to help improve connectivity between physicians not in the same locale, increase efficiency and provide better access to vital information used in a medical and surgical setting. The device has clear teaching implications and will enable academic physicians to disseminate information to more students and in situations not previously possible. As the device evolves its potential to do more will likely develop further. It is important to assess the impact of this rapidly growing field on patient sentiment and wellbeing. As this is a very new device, very few studies have been done to assess its application in Medicine and specifically orthopaedic surgery. So far only very specific and small studies have been done with regard to immunochromatographic analysis, pharmacology, forensic medicine and Parkinson's disease. The investigators are aiming to assess the applications and patient perspective of this device on a much larger scale. The investigators feel this technology and its future offspring could be polarizing with regard to patient response. This could be an important element to consider in the future development of its clinical applications.

There are no direct medical risks to the patient. No decisions regarding patient care will be dependent on the device.

Study Objective Primary question: What is the patient's level of acceptance and response to this new technology? Secondary question: From a doctor's perspective, how effective is this new tool in the Orthopaedic clinical setting?

Design Patients seen in the Orthopaedic Trauma clinic will be asked to consent for potential video/picture recording using the Google Glass device during their visit with the orthopaedic surgeon or resident. Eligible patients will be assigned to one of two consulting rooms: one with the Google Glass device, one without.

Patients will therefore have a 50.50 chance of encountering the Google Glass.

Any images or videos taken will not show the patients face, all measures will be taken to ensure confidentiality. Both groups will be asked to complete a small survey on a locked password protected iPad after their visit so as to record their acceptability of this new technology in a clinical setting. Participants that experienced the device will also be required to comment on their experience. The device user (surgeon/resident) will also complete a survey so as to record their experience using the hands free camera and recording device.

The information gathered will be saved on a password protected drive and will be used for discussion and analysis between the investigators to help develop the potential future teaching and clinical applications of the device.

ELIGIBILITY:
Inclusion Criteria:

* All patients seen in the Montreal general Hospital (MGH) - Orthopaedic Trauma Clinic and capable of reading French or English.

Exclusion Criteria:

* All patients that have cognitive impairment or language difficulties that would impede completion of the survey will be excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2014-08; Primary Completion 2018-05-30 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Patient Evaluation Survey | Day one

SECONDARY OUTCOMES:
Surgeon Evaluation Survey | Day one

CONTACTS AND LOCATIONS:
Overall Officials: Edward J Harvey, MDCM FRCSC, Principal Investigator — RI-MUHC
Locations (1):
- Montreal General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No